CLINICAL TRIAL: NCT02965651
Title: A Randomized Controlled Trial of A Virtual Patient Advocate System: "Go to Gabby" for Health and Wellness Information
Brief Title: Engaging Women With the Gabby System to Deliver Multiple Health-Related Behavioral Changes: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Paula Gardiner, Associate Professor, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-30418
Record Dates: First submitted 2016-11-07; First posted 2016-11-17 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Stress, Emotional
Keywords: embodied conversational agent; virtual patient agent; meditation; mindfulness based stress reduction; nutrition
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECA System (Experimental): Access to website and virtual patient advocate
  Interventions: Behavioral: ECA System
- Standard of Care (No Intervention): Patient information sheets and meditation CD

INTERVENTIONS:
Behavioral: ECA System — The ECA system, named "Gabby", included content pertaining to stress management, nutrition and physical activity as well as dialogue scripts and media such as meditations. The scripts included motivational interviewing dialogue: dialogue to simulate shared decision making interactions and additional longitudinal interaction using techniques such as "goal setting," "problem solving," "tips," and "homework". Gabby was available on a web browser through a username and secure password login.
  Arms: ECA System

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the feasibility of introducing an innovative eHealth technology, the Embodied Conversational Agent (ECA), to diverse women from an urban outpatient setting.

DETAILED DESCRIPTION:
This trial focuses on using an embodied conversational agent (ECA) named Gabby to teach healthy lifestyle behaviors (healthy eating, exercise, stress reduction). This feasibility randomized control trial will include 70 women in the outpatient setting (35 intervention and 35 controls). The control group will receive usual care (patient information sheets on healthy eating, exercise, stress reduction and a CD with meditation, body scan, and mindful yoga).

The ECA is an animated conversational character who simulates face-to-face interaction with a patient. During the intervention, the ECA talks using synthetic speech and synchronized animation; patients "talk" by clicking what they want to say using a computer's mouse. The ECA delivers information and experiential on stress (principles of mindfulness based stress reduction such as: meditation, yoga, body scan), nutrition, and exercise.

If participants are randomized to the intervention, a research assistant (RA) will teach the subject how to use the ECA workstation. The ECA will review with the patients their nutrition, stress, exercise, using the ECA workstation which will also be programmed with the subject's baseline information (e.g., name, age). Subjects will be asked to log onto the system once a day and interact with the system for as long as they wish.

Prior to the midpoint survey, participants will receive a reminder phone call/email. At 14 days, the RA will survey all participants regarding satisfaction with either the ECA or the paper handouts, and whether or not they are adhering to the lifestyle modification recommendations. This will be conducted either by email, phone or in person.

Prior to the end of the 30 day study participation, the RA will call or email to schedule a visit to complete the post intervention questionnaire. The RA will call/email 1-2 days before the final study visit to remind the participant.

The RA will conduct the post intervention interview in person or by phone. All participants received compensation for completion of surveys.

Control Group: The control subjects will receive usual care (patient information sheets on stress, nutrition and exercise and a CD). The RA will administer the same baseline, mid-point and final surveys to the control participants.

The investigators do not know, however, whether health information technology can be used effectively to deliver information on exercise, nutrition and stress in the outpatient setting. This study will add new information to the viability of using the ECA in women in the outpatient setting compared to patient information sheets.

ELIGIBILITY:
Inclusion Criteria:

* English fluency sufficient to follow treatment instructions and answer survey questions
* Access to a telephone (landline, cellular phone)
* Access to a computer/laptop with internet/Wi-Fi access

Exclusion Criteria:

* Known or planned pregnancy
* Mental health or substance abuse problems that would bar completion of study
* Refusal of consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of people recruited | 1 year
Number of participants who completed the study | 1 month
Number of participants whom outcome data can be collected | 1 month
Number of participants who were racial minorities (non-white) | 1 month
Participant satisfaction with either treatment arm | 1 month
  Likert scale of 1-7 (1=not satisfied, 7=very satisfied)

SECONDARY OUTCOMES:
Age | 1 month
Race | 1 month
Ethnicity | 1 month
Education Level | 1 month
Work Status | 1 month
Income Level | 1 month
BMI | 1 month
  Height (ft) and weight (lbs)
Health Conditions | 1 month
  Self-reported; cross-checked with medical records
Medication Use | 1 month
  Self-reported; cross-checked with medical records
Smoking Status | 1 month
Pain Levels | 1 month
  Pain scale of 0-10 (0=no pain, 10=worst possible pain)
Depression | 1 month
  Patient Health Questionnaire - 9 items
Stress Level | 1 month
  Perceived Stress Scale - 4 items
Dietary Patterns | 1 month
  Nutrition Survey
Food Access | 1 month
  Household Food Insecurity Access Scale
Physical Activity | 1 month
  Stanford Patient Education Research Center Exercise Behaviors
Number of Logins into the ECA | 1 month
  Intervention users only
Duration of ECA Use | 1 month
  Intervention users only (minutes)
Technical issues | 1 month
  Intervention users only

CONTACTS AND LOCATIONS:
Overall Officials: Paula Gardiner, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gardiner P, Hempstead MB, Ring L, Bickmore T, Yinusa-Nyahkoon L, Tran H, Paasche-Orlow M, Damus K, Jack B. Reaching women through health information technology: the Gabby preconception care system. Am J Health Promot. 2013 Jan-Feb;27(3 Suppl):eS11-20. doi: 10.4278/ajhp.1200113-QUAN-18. PMID 23286652